CLINICAL TRIAL: NCT02808169
Title: Radlinik GPS Provide a Valid Intra-operative Assessment of Acetabular Inclination and Anteversion
Brief Title: Radlink GPS Provide a Valid Intra-operative Assessment of Acetabular Inclination and Anteversion
Status: Completed | Type: Observational
Sponsor: Barrett, William, M.D. (Individual)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Principal Investigator, William Barrett, M.D., William P. Barrett, MD, Barrett, William, M.D.
Other Study IDs: 20151031
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Implant Position in Total Hip Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluate the accuracy of Radlink System in determining acetabular cup placement and limb length evaluation during Anterior hip replacement as measured intraoperative with C-Arm visualization and confirmed with digital x-ray at 4-6 weeks postoperatively.

DETAILED DESCRIPTION:
Evaluate the accuracy of Radlink System in determining acetabular cup placement and limb length evaluation during Anterior hip replacement as measured intraoperative with C-Arm visualization and confirmed with digital x-ray at 4-6 weeks postoperatively.

GPS may improve total hip replacement by allowing surgeons to measure the exact position of components placed during surgery and there is a question whether RADLINK helps surgeons place the acetabular cup (the part that goes into the hip bone) component in a precise position. The objective of the study is to determine whether GPS gives surgeons reliable, valid information about the orientation of the cup component. The surgeons need to collect data to help clarify this issue.

ELIGIBILITY:
Inclusion Criteria:

* Both: both female and male participants are being studied.
* Minimum Age: Age of participants is between 20 years - 75 years.
* Accepts: Persons who are in need of a total hip replacement

Exclusion Critieria:

* Has an existing condition that would compromise participation
* Had previous surgery on affected hip

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient under going total hip replacement
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2016-08-08 (Actual); Study Completion 2016-08-08 (Actual)

PRIMARY OUTCOMES:
Comparison of intra-op values for acetabular inclination and ante version, limb length using Radlink with those obtained and 4-8 weeks postop digital films. | 4-8 weeks

SECONDARY OUTCOMES:
Accuracy of cup placement/limb length with Radlink to a predetermined value and what surgeon obtains with Radlink guidance. | 4-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Barrett, MD, Principal Investigator — VOA Research Foundation
Locations (1):
- VOA Research Foundation, Renton, Washington, United States